CLINICAL TRIAL: NCT03900273
Title: Development of Novel Measures of Cognition and Function for Alzheimer's Disease Prevention Trials
Brief Title: Development of Novel Measures for Alzheimer's Disease Prevention Trials
Acronym: NoMAD
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The NYSPI site is currently paused and has been paused since an institutional pause on human subjects research began in June 2023.
  The U.S. Department of HHS Office of Human Research Protections (OHRP) issued a pause on human subjects research.
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Columbia University (Other); University of Southern California (Other); Feinstein Institute for Medical Research (Other); University of Miami (Other)
Responsible Party: Principal Investigator, Terry Goldberg, Professor of Medical Psychology, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 7672
Record Dates: First submitted 2019-03-15; First posted 2019-04-03 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Healthy Participants
Keywords: Alzheimer's disease; Neuropsychological Testing; Healthy Older Individuals; Psychometrics; Prevention; Clinical Trial
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel measures of cognition and everyday function (Experimental): No Practice Effects (NPE) cognitive battery
  Miami Computerized Functional Assessment Scale (CFAS)
  Participants will receive three serial assessments of the NPE and CFAS over a one year period. Assessments will take place at baseline, week 12, and week 52.
  Interventions: Other: No Practice Effects (NPE) cognitive battery, and Miami Computerized Functional Assessment Scale (CFAS)
- Established measures of cognition and everyday function (Active Comparator): Preclinical Alzheimer's Cognitive Composite (PACC)
  Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog)
  Functional Assessment Questionnaire (FAQ).
  Participants will receive three serial assessments of the PACC, ADAS-Cog and FAQ over a one year period.
  Assessments will take place at baseline, week 12, and week 52.
  Interventions: Other: Preclinical Alzheimer's Cognitive Composite (PACC), Alzheimer's Disease Assessment Scale-Cognitive Scale (ADAS-Cog), and Functional Assessment Questionnaire (FAQ)

INTERVENTIONS:
Other: No Practice Effects (NPE) cognitive battery, and Miami Computerized Functional Assessment Scale (CFAS) — Novel measures of Cognitive and Everyday function
  Arms: Novel measures of cognition and everyday function
Other: Preclinical Alzheimer's Cognitive Composite (PACC), Alzheimer's Disease Assessment Scale-Cognitive Scale (ADAS-Cog), and Functional Assessment Questionnaire (FAQ) — Established measures of Cognitive and Everyday Function
  Arms: Established measures of cognition and everyday function

SUMMARY:
This protocol focuses on novel measures of cognition and everyday function that have robust psychometrics and reduced practiced effects. They will be deployed in a parallel group study in which participants are randomized to assessment type (novel vs established) and receive serial assessments over a one year period in order to highlight contrasts between novel and established measures.

DETAILED DESCRIPTION:
This protocol has the goal of validating novel cognitive and everyday functional measures that have sharply attenuated practice effects and are not prone to ceiling effects for use in preclinical Alzheimer's disease (AD) trials in which participants are cognitively within normal limits. To implement this, we will conduct an innovative parallel group study in which 400 healthy, non-cognitively impaired older subjects are randomized to one of two groups based on assessment type (novel instruments vs. established) and receive three serial assessments over a one year period. Novel cognitive measures include tests of executive function, episodic memory, and processing speed combined into a single composite. Novel functional measures involve computerized performance based, ecologically relevant instrumental activities. We will compare our novel No Practice Effects (NPE) cognitive battery and Miami Computerized Functional Assessment Scale (CFAS) against established measures that include the ADAS-COG in order to determine which battery (novel or established) has better psychometric properties and is less sensitive to practice effects in this clinical trials structure.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking participants, ages 60-85 years
2. MMSE score of 24 or greater
3. Logical Memory II score of 9 or greater for subjects with 16 or more years of education, 5 or more for subjects with 8-15 years of education, and 3 or greater for subjects with 0-7 years of education
4. Presence of subjective memory complaints not exclusionary
5. A family member or other individual who is in contact with the subject and consents to serve as informant during the study.

Exclusion Criteria:

1. Diagnosis of stroke or excessive risk of CVD
2. Neurologic disease including movement disorders, MS, epilepsy, and TBI (with greater than 15 min loss of consciousness)
3. Untreated diabetes
4. Current DSM-5 Axis I psychiatric diagnosis of schizophrenia schizoaffective disorder or bipolar disorder; current major depression as determined by a Geriatric Depression Scale score of greater than 5. Current alcohol or substance use disorder
5. Active treatment of cancer
6. MMSE score below 24 and Logical Memory below 9 for subjects with 16 or more years of education, 5 for subjects with 8-15 years of education, and 3 for subjects with 0-7 years of education
7. Females who are pre-menopausal and are pregnant.
8. Use of antidepressants with large anticholinergic properties will be excluded. These include: amitriptyline, amoxapine, clomipramine, desipramine, doxepin, imipramine, isocarboxazide, lithium, maprotiline, mirtazapine, nortriptyline, tranylcypromine trimipramine, and phenelzine.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-02-25 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Computerized Functional Assessment Scale (CFAS). | Baseline to Week 52; change in score will be assessed
  Novel computerized measure of everyday function. Testing format is a set of simulations (ATM use, Kiosk ticket purchase , Prescription refill , and Doctor's visit ). We will construct a z score based on the "rate" measure which accounts for both speed and accuracy. Higher scores suggest greater cognitive function while lower scores indicate greater cognitive impairment.
No Practice Effect (NPE) Cognitive Battery. | Baseline to Week 52; change in score will be assessed
  Novel measure of cognitive function. Scores can be age-adjusted by decade. The majority of the subtests ( including tests of Cognitive Control/Executive Processes, Working Memory,Speed of Processing,Verbal Fluency and Episodic Memory)are computerized or partially computerized. All tests have three equivalent alternate forms. We will construct a z-score averaged composite based on scores of the subtests at baseline. Higher scores suggest greater cognitive function while lower scores indicate greater cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Terry E. Goldberg, Ph.D., Principal Investigator — Columbia University Medical Center/ New York State Psychiatric Institute
Locations (4):
- United States (4):
  - University of Southern California, Los Angeles, California
  - University of Miami, Miami, Florida
  - The Feinstein Institute for Medical Research, Manhasset, New York
  - New York State Psychiatric Institute, New York, New York

REFERENCES:
- [Background] Goldberg TE, Harvey PD, Wesnes KA, Snyder PJ, Schneider LS. Practice effects due to serial cognitive assessment: Implications for preclinical Alzheimer's disease randomized controlled trials. Alzheimers Dement (Amst). 2015 Mar 29;1(1):103-11. doi: 10.1016/j.dadm.2014.11.003. eCollection 2015 Mar. PMID 27239497
- [Derived] Bell SA, Cohen HR, Lee S, Kim H, Ciarleglio A, Andrews H, Rivera AM, Igwe K, Brickman AM, Devanand DP, Harvey PD, Schneider LS, Goldberg TE. Development of novel measures for Alzheimer's disease prevention trials (NoMAD). Contemp Clin Trials. 2021 Jul;106:106425. doi: 10.1016/j.cct.2021.106425. Epub 2021 Apr 30. PMID 33933666